CLINICAL TRIAL: NCT01602068
Title: A Prospective, Multi-Center, Randomized, Double-Masked, Negative-Controlled Clinical Trial Designed to Compare the Safety and Efficacy of EGP-437 (Dexamethasone Phosphate Ophthalmic Solution) Delivered by EyeGate® II Iontophoresis to Placebo in Patients Undergoing Cataract Surgery With Implantation of a Posterior Chamber Intraocular Lens
Brief Title: Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Delivery Prior to Implantation of a Posterior Chamber IOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-005
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Cataract
Keywords: Iontophoresis; Cataract Surgery; Ophthalmology; Posterior Chamber Intraocular Lens Implant
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone Phosphate Ophthalmic (Experimental): Dexamethasone Phosphate Ophthalmic: (40 mg/mL) solution delivered by ocular iontophoresis consisting of 4.0 mA-min at 1.5 mA on Day -1 (the day before cataract surgery)
  Interventions: Drug: Dexamethasone Phosphate Ophthalmic
- 100 mM Sodium Citrate Buffer (Placebo Comparator): Placebo (100 mM sodium citrate buffer solution) delivered by ocular iontophoresis consisting of 4.0 mA-min at 1.5 mA on Day -1 (the day before cataract surgery)
  Interventions: Drug: 100 mM Sodium Citrate Buffer

INTERVENTIONS:
Drug: Dexamethasone Phosphate Ophthalmic — Transcleral iontophoresis delivery of EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis)
  Other Names: Active arm, Arm 1
  Arms: Dexamethasone Phosphate Ophthalmic
Drug: 100 mM Sodium Citrate Buffer — Transcleral iontophoresis delivery of 100 mM sodium citrate buffer solution
  Other Names: In-active control arm, Arm 2
  Arms: 100 mM Sodium Citrate Buffer

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ocular iontophoresis with dexamethasone phosphate ophthalmic solution EGP-437 using the EyeGate® II Drug Delivery System (EGDS) compared to placebo in patients undergoing cataract surgery with implantation of a posterior chamber intraocular lens.

DETAILED DESCRIPTION:
Phase 2, proof-of-concept (POC) clinical trial designed to evaluate the safety and efficacy of ocular iontophoretic delivery of dexamethasone phosphate ophthalmic solution compared to ocular iontophoresis with a placebo (100 mM citrate buffer of pH 5.7) in patients planning to have cataract surgery with implantation of a posterior chamber intraocular lens (IOL). The population studied was comprised of males and females scheduled for unilateral cataract surgery with implantation of a posterior chamber IOL. Eligible patients were enrolled into the study and were randomized on Day 1 in a 1:1 ratio into one of the following two treatment arms. Treatments were administered on the day prior (Day -1) to cataract surgery (Day 0). Subjects were scheduled to return to the clinic on Days 1, 7, 14, and 28. All subjects were scheduled to exit the study on Day 28. Subjects were asked to complete a daily pain score assessment questionnaire for the first 14 days post-surgery (Days 0 - 14).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing unilateral cataract extraction and implantation of a monofocal IOL (at the time of enrollment)
* Male or female 18 years or older
* Receive, understand, and sign a copy of the written informed consent form
* Be able to return for all study visits and willing to comply with all study-related instructions

Exclusion Criteria:

* Subjects not meeting the inclusion criteria
* Subjects being implanted with a multifocal IOL
* Ocular surgery of any kind in the study eye within 6 months prior to baseline visit
* Cataract surgery on the fellow eye within 6 weeks, including 2 weeks without topical ocular medication, prior to baseline visit
* Scheduled for surgery in the fellow eye within the study period
* Have anterior chamber inflammation as measured by slit lamp examination at baseline. Anterior chamber cell and/or flare grade > 0
* Have used any topical ocular medication in either eye, other than tear substitute for dry eye, at least 2 weeks prior to baseline visit
* Have IOP ≥ 25 mmHg at baseline, a history of glaucoma, or require ocular anti-hypertensive medications
* Be known corticosteroid intraocular pressure responder in either eye
* Have used topical corticosteroid or NSAID treatment in either eye ≤ 48 hours prior to baseline visit
* Systemic administration of corticosteroid within the past 14 days prior to baseline visit
* Have received intravitreal, sub-Tenon's, or any periocular corticosteroid treatment in either eye within the past 6 months prior to baseline visit
* Have open wounds/ skin disease on the forehead area where the iontophoresis return electrode will be applied
* Have severe lesions of the eyelids or the ocular surface impeding the application of the iontophoresis applicator
* Have blepharospasm, blepharophimosis, or other eyelid anatomic variations precluding the placement of the iontophoresis applicator
* Have significant Fuch's Corneal Dystrophy
* Have known allergy to dexamethasone or dexamethasone phosphate or any medication to be used in this study
* Have history or diagnosis of ocular herpes, corneal lesion of suspected herpetic origin
* Have optic neuritis of any origin
* Have clinically suspected or confirmed central nervous system or ocular lymphoma
* Have active hyphema, pars planitis, choroiditis, Behçet's disease, clinically significant macular edema, toxoplasmosis scar, or vitreous hemorrhage
* Have severe/serious ocular pathology or medical condition which may preclude study completion
* History of HIV/AIDS
* Have pacemaker and/or any other electrical sensitive support system
* Be pregnant or lactating female, or female of childbearing age and using inadequate birth control method
* Have participated in another investigational device or drug study within 30 days of baseline visit
* Have already participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, M.D., Principal Investigator — Center For Excellence In Eye Care
Locations (3):
- United States (3):
  - Site 501, Miami, Florida
  - Site 503, Tamarac, Florida
  - Site 502, Washington, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female patients at least 12 years of age and undergoing unilateral cataract surgery with implantation of a posterior chamber IOL could be screened
Pre-assignment Details: 1:1 randomization
Groups:
- Dexamethasone Phosphate Ophthalmic: Dexamethasone Phosphate Ophthalmic: (40 mg/mL) solution delivered by transcleral iontophoresis consisting of 4.0 mA-min at 1.5 mA on Day -1 (the day before cataract surgery)
- 100 mM Sodium Citrate Buffer: Placebo (100 mM sodium citrate buffer solution) delivered by transcleral iontophoresis consisting of 4.0 mA-min at 1.5 mA on Day -1 (the day before cataract surgery)
Period: Overall Study
Arm/Group | Dexamethasone Phosphate Ophthalmic | 100 mM Sodium Citrate Buffer
Started | 23 (Day before surgery) | 22 (Day before surgery)
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients planning to undergo a unilateral, posterior IOL.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Phosphate Ophthalmic | 100 mM Sodium Citrate Buffer | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Full Range); unit: years] | 59 [12 to 81] | 65 [50 to 80] | 62 [12 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With AC Cell Count of Zero on Day 7
Description: Percentage of patients with anterior chamber (AC) cell count of zero on Day 7 as compared between the active and placebo groups
Time Frame: At Day 7 (plus or minus two days) following the study treatment
Population: This was an exploratory study and therefore a number of efficacy and safety parameters were evaluated. In all measures there was no significant difference between the active and non-active arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Phosphate Ophthalmic | 100 mM Sodium Citrate Buffer
Number analyzed (Participants) | 23 | 22
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: AEs were collected from the point that the ICF was signed. All AEs until the last day of the study, through resolution, stabilization, or at least 30 days after treatment, whichever occurs first.
Arm/Group | Dexamethasone Phosphate Ophthalmic | 100 mM Sodium Citrate Buffer
Serious Adverse Events (participants affected / at risk) | 0/23 | 3/22
Other Adverse Events (participants affected / at risk) | 21/23 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Phosphate Ophthalmic (N=23) | 100 mM Sodium Citrate Buffer (N=22)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related. Between Visits 5 & 6.
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related. Between Visits 5 & 6.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related. Between Visits 5 & 6.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Phosphate Ophthalmic (N=23) | 100 mM Sodium Citrate Buffer (N=22)
Ocular AE (Eye disorders) | 21 (84) | 20 (70) — In Study eye

LIMITATIONS AND CAVEATS:
The surgical procedure eliminates or washes out any remaining study drug product from the ocular tissue which becomes inflamed post-surgery. Exploratory study with multiple efficacy & safety parameters were evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other